CLINICAL TRIAL: NCT01500486
Title: Observational Study to Assess Ease of Use, Acceptability and Preference of Norditropin NordiFlex® With NordiFlex PenMate™ in Subjects on Prescribed Growth Hormone Therapy
Brief Title: Observational Study of Norditropin NordiFlex® With NordiFlex PenMate™
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GH-3717
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Growth Hormone Disorder; Growth Hormone Deficiency in Children; Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PenMate device
  Interventions: Device: NordiFlex PenMate™

INTERVENTIONS:
Device: NordiFlex PenMate™ — Subjects whom will be offered growth hormone (Norditropin NordiFlex®) on prescription as part of normal clinical practice will be asked to evaluate the NordiFlex PenMate™ device.

SUMMARY:
This study is conducted in Europe. The aim of this study is to evaluate ease of injection of growth hormone in patients using Norditropin NordiFlex® with NordiFlex PenMate™. Convenience and tolerability of NordiFlex PenMate™ - an automatic injection and a needle hiding device - is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* After the physician decision has been made to use Norditropin Nordiflex® growth hormone therapy in accordance with the locally approved labelling, any subject is eligible for the study, including newly diagnosed subjects who have never received growth hormone therapy before and subjects who were treated with the other growth hormone products (with exclusion of patients who received previously Norditropin Nordiflex®) and need to be switched to a new product. The selection of the subjects will be at the discretion of the individual physician

Exclusion Criteria:

* Contraindications to Norditropin® growth hormone therapy
* Subjects who have received Norditropin NordiFlex® prior to this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects from secondary care physicians who prescribe growth hormone will be included in the study. Children who are available for Norditropin® treatment in accordance with the labelling will be included in the study: Newly-diagnosed subjects who have never received growth hormone therapy before and subjects in whom physician identifies a need for switch to another growth hormone preparation
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects that find growth hormone injection using Norditropin Nordiflex® with NordiFlex PenMate™ very easy or easy as assessed by patient/parent questionnaire | Week 12

SECONDARY OUTCOMES:
Ease of teaching how to use Norditropin Nordiflex® with NordiFlex PenMate™ as assessed by nurse questionnaires | Week 0
Patient/parent overall acceptance of Norditropin Nordiflex® with NordiFlex PenMate™ as assessed by questionnaire | Week 12
Compliance to treatment as assessed by patient/parent diary | Week 12
Evaluation of tolerability, when using Norditropin Nordiflex® with NordiFlex PenMate™, by collecting Adverse Drug Reactions (ADRs), Serious Adverse Drug Reactions (SADRs) and clinical technical complaints | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- Novo Nordisk Investigational Site, Mainz, Germany
- Novo Nordisk Investigational Site, Alphen aan den Rijn, Netherlands
- Novo Nordisk Investigational Site, Malmo, Sweden

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com